CLINICAL TRIAL: NCT04156334
Title: The Effect of Two Local Anaesthesia Techniques on the Paediatric Patient's Recovery After Dental Treatment in General Anaesthesia
Brief Title: The Effect of Local Anaesthesia Technique on the Recovery After Dental Treatment in General Anaesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019/01
Record Dates: First submitted 2019-09-12; First posted 2019-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Anesthesia, Local

STUDY DESIGN:
Intervention Model Description: The double-blinded prospective randomised study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Concealed randomisation table where patients will be consecutively assigned. Every patient will be given a number according to the randomisation table and the study group inclusion will not be revealed to the investigator or patients until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- computer-controlled intraosseous anaesthesia (Experimental): Patients will receive the local anaesthetic using computer-controlled intraosseous anaesthesia (Quicksleeper 5) before the tooth extraction in general anaesthesia.
  Interventions: Procedure: Extraction of teeth in general anaesthesia using either computer-controlled intraosseous anesthesia device or carpule for local anaesthesia
- infiltrative or conductive local anaesthesia (Experimental): Patients will receive a local anaesthetic using carpule before the tooth extraction in general anaesthesia.
  Interventions: Procedure: Extraction of teeth in general anaesthesia using either computer-controlled intraosseous anesthesia device or carpule for local anaesthesia

INTERVENTIONS:
Procedure: Extraction of teeth in general anaesthesia using either computer-controlled intraosseous anesthesia device or carpule for local anaesthesia — QuickSleeper 5 with DHT needles or carpule with periapical/nerve block needles will be used to administer local anaesthetic before teeth extraction in general anaesthesia.

SUMMARY:
Use of local anaesthesia during full mouth dental rehabilitation under general anaesthesia is an everyday practice. It enables better control of the post-extraction bleeding and better control of physiological responses. Postoperative numbness and lip and cheek biting can be an undesired side effect. With our research, we aim to compare two different types of local anaesthesia in relation to postoperative side effects. We also aim to assess the oral health-related quality of life after treatment in general anaesthesia to enlighten how full mouth rehabilitation affects a child's life.

DETAILED DESCRIPTION:
Dental treatment of children under general anaesthesia (GA) is intended for children who, for one reason or another, are unable to participate in the outpatient clinic.

When extracting teeth in GA, local anaesthetics (LA) are regularly applied to control bleeding, reduce postoperative sensitivity, and to better control vital functions. The side effects of LA can be the patient's irritation due to not understanding the postoperative numbness and lip and cheek biting.

The aim of our study is to determine if there is a difference between the two types of local anaesthesia (computer-controlled intraosseous anaesthesia and classical local/conductive anaesthesia) in the frequency and extent of the occurrence of side effects postoperatively.

The research data would help establish a better dental extraction protocol for children under GA, which would allow for less postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

- Paediatric patients intended for dental treatment in general anaesthesia

Exclusion Criteria:

* Patients who can not express feelings adequately,
* patients where there will not be any teeth extracted,
* patients whose parents do not want to participate in the study

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Pain scores before and over 48 hours after tooth extraction in general anaesthesia in the two study groups using The Children's Hospital of Eastern Ontario Pain over Scale (CHEOPS) | an average 51 hours (monitoring of pain will be performed one hour before the general anesthesia treatment, 2 hours after treatment, 12 hours after treatment, 24 and 48 hours after treatment
  Monitoring's the pain with CHEOPS which evaluates crying, face expression, speech, body movement, touching of the painful area and leg movement. Each category has specific points according to the level of behaviour. Points are added and final scores range between 4-13 points. The number of scores at different measuring points before and over 48 hours after treatment will be compared between the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Rok Gašperšič, Phd, Study Chair — University of Ljubljana
Locations (1):
- University medical centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No
non

REFERENCES:
- [Result] Patini R, Staderini E, Cantiani M, Camodeca A, Guglielmi F, Gallenzi P. Dental anaesthesia for children - effects of a computer-controlled delivery system on pain and heart rate: a randomised clinical trial. Br J Oral Maxillofac Surg. 2018 Oct;56(8):744-749. doi: 10.1016/j.bjoms.2018.08.006. Epub 2018 Aug 22. PMID 30143396
- [Result] Townsend JA, Ganzberg S, Thikkurissy S. The effect of local anesthetic on quality of recovery characteristics following dental rehabilitation under general anesthesia in children. Anesth Prog. 2009 Winter;56(4):115-22. doi: 10.2344/0003-3006-56.4.115. PMID 20020791